CLINICAL TRIAL: NCT04899791
Title: Positive Effects of Daily Consumption of Bread Enriched With Hydroxytyrosol on the Results of a 12-week Dietary Intervention on Subjects With Type 2 Diabetes Mellitus and Overweight/ Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vaios T. Karathanos, Professor of Food Engineering and Physical Chemistry, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Harokopio_EnrichedBread
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheat bread enriched with hydroxytyrosol (Experimental)
  Interventions: Other: Wheat bread enriched with hydroxytyrosol
- Wheat bread (Active Comparator)
  Interventions: Other: Wheat bread

INTERVENTIONS:
Other: Wheat bread enriched with hydroxytyrosol — Wheat bread enriched with hydroxytyrosol
  Arms: Wheat bread enriched with hydroxytyrosol
Other: Wheat bread — Wheat bread
  Arms: Wheat bread

SUMMARY:
Hydroxytyrosol is a phenolic compound drawn from the olive tree and its leaves as a by-product obtained from the manufacturing of olive oil and has antioxidant and antidiabetic effects. The use of HT extract in food products is a good strategy to improve their nutritional quality. However, this extract has a strong odour and flavour, so it is important to be encapsulated for the odour and flavour to be covered up. The purpose of the study is to investigate the effects of regular consumption of bread enriched with HT on biochemical parameters (blood glucose and cholesterol levels).

DETAILED DESCRIPTION:
Subjects with type 2 diabetes mellitus and overweight/ obesity will participate in the present study. They will follow a 12-week energy-restricted dietary intervention supplemented with a certain amount of bread enriched with hydroxytyrosol. The effects of the dietary intervention on biochemical parameters (blood glucose and cholesterol levels) and body weight reduction will be examined.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* bmi : 25-40 kg/ m-2
* normal exercise and dietary habits
* weight stable for at least 3 months before enrollment

Exclusion Criteria:

* HbA1C > 8.5%
* pregnancy
* chronic medical illness
* regular intense exercise
* alcohol consumption (> 2 drinks/day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C levels | 12 weeks
  Change in HbA1C levels after energy-restricted dietary intervention with wheat bread enriched with hydroxytyrosol compared to conventional wheat bread
Change in blood cholesterol levels | 12 weeks
  Change in blood cholesterol levels after energy-restricted dietary intervention with wheat bread enriched with hydroxytyrosol compared to conventional wheat bread

SECONDARY OUTCOMES:
Change in body weight | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Laiko General Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Attica
  - Laiko General Hospital of Athens, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Binou P, Stergiou A, Kosta O, Tentolouris N, Karathanos VT. Positive contribution of hydroxytyrosol-enriched wheat bread to HbA1c levels, lipid profile, markers of inflammation and body weight in subjects with overweight/obesity and type 2 diabetes mellitus. Eur J Nutr. 2023 Aug;62(5):2165-2176. doi: 10.1007/s00394-023-03133-9. Epub 2023 Apr 5. PMID 37017765